CLINICAL TRIAL: NCT02735226
Title: Shanghai Stroke Service System
Brief Title: Stroke Prevention and Treatment System in Shanghai: a Network of Public Healthcare of Stroke
Acronym: SSSS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Stroke Service System (Other)
Collaborators: Huashan Hospital (Other); Shanghai Zhongshan Hospital (Other); Ruijin Hospital (Other); theTenth People's Hospital (Unknown); the Sixth People's Hospital (Ambiguous); RenJi Hospital (Other); ShuGuang Hospital (Other); Dongfang Hospital Beijing University of Chinese Medicine (Other); Changzheng Hospital (Unknown); Changhai Hospital (Other); the Ninth People's Hospital (Unknown)
Responsible Party: Principal Investigator, Qiang Dong, Director of Shanghai Stroke Service system, Shanghai Stroke Service System
Other Study IDs: Shanghai Stroke Service System
Record Dates: First submitted 2016-03-31; First posted 2016-04-12 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Stroke
Keywords: stroke; Shanghai Healthcare; Healthcare Quality, Access, and Evaluation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Acute Stroke patient: Patients who are presented to hospital within 7days from onset. The key measurement of clinical quality controlled in patients with acute stroke managment and inhouse stroke care were record automatically
  Interventions: Other: stroke network and policy intervention

INTERVENTIONS:
Other: stroke network and policy intervention — Shanghai stroke service and network contributes to update the ability of stroke care of comprehensive and primary stroke center,to improve radiation ability of comprehensive stroke centers and try to form a close relationship between comprehensive stroke centers and its primary stroke centers.

SUMMARY:
The Shanghai Stroke Service System（4S） has been established as the network of stroke care in greater Shanghai metropolitan area. The system includes 11 territorial-care hospitals and their comprehensive stroke unites that provide 24h/7day acute stroke care to a population of 40 million in Shanghai. The System comprised of two consecutive phases, the acute phase that emphasized on providing thrombolysis, and the in-hospital phase that concentrated on the effort of recovery and secondary stroke prevention. The novel electronic data aquisition system provides the contiguous data of clinical care of stroke patients from the acute phase of management to inpatient rehabilitation. This system has been implemented and maintained as an ongoing quality of stroke care project that monitored the process of routine stroke care in Shanghai. It is funded by the Shanghai Municipal Commission of Health and Family Planning. Our analysis of the project was approved by the Ethics Committee, which agreed that no written informed consents were needed since the study only was consisted of a population-based retrospective data analysis.

DETAILED DESCRIPTION:
The goal of Shanghai stroke service system is to promote and facilitate high quality standardized stroke care in Shanghai area. The 11 hospitals involved are committed to provide the best stroke care to their patients. This quality goal consists of two parts: the acute phase of stroke care and the subsequent care during the hospitalization. To accomplish this goal, each hospital has organized a multidisciplinary stroke team that will address day-to-day stroke care. Each hospital provides prioritized neuroimaging service to patients with acute stroke 24hr per day, 7days per week. A stroke neurologist is on site 24hr per day, 7 days per week in each hospital. This team will follow the guidelines to carry out standardized secondary stroke prevention once the patient has been admitted.

The stroke clinical pathway is available on line in computers of each hospital. This pathway can be accessed from hospital computers, or from outside.

Stroke team members in each hospital obtained and entered all data on each stroke patient: demographics, stroke onset time, onset to thrombolytic time, presenting NIHSS, timing of diagnostic procedures, treatment strategies, performance of quality measures, comorbidities, in-hospital mortality, etc. These data are contained in a three-page form, which are embedded in the electronic health record of each patient.

If ICD-10 stroke codes were entered as the primary discharge diagnoses, the electronic health record systems would not allow the discharge of the patient until all required documentation has been completed. The EHR would not allow for any empty fields before it could be closed. Data quality was assured by automatic feasibility checks. The novel electronic data acquisition system provides the continuous clinical care data on all stroke patients from their acute management phase to inpatient rehabilitation or discharge.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* primary diagnosis as acute stroke or TIA within 7 days from onset
* admitted in stroke unit.

Exclusion Criteria:

* child or teenager younger than 18 years old
* woman with pregnant
* outpatient
* any other reason that patient cannot be admitted for secondary prevention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with acute stroke are admitted to these 11 hospital in Shanghai for secondary prevention.
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2014-01; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
The acute stroke service and treatment provided in Shanghai area | 5 years
  The phase of acute stroke therapy. Under this category, the acute stroke care specific quality measurement items are:
  Stroke onset to hospital ER Time
  Door to CT Time
  Door to seen by a doctor Time
  Door to IV TPA Time
  Door to groin puncture time for IA therapy
  Door to admission to a hospital bed Time
The secondary prevention of stroke provided after discharge in Shanghai area | 5 years
  2. Secondary stroke prevention prescribed.
  Antithrombotics prescribed
  Swallowing evaluation performed before oral feeding starts
  DVT prophylaxis prescribed
  Anticoagulation for atrial fibrillation prescribed
  Brain imaging including vascular imaging performed
  Stroke education provided
  Educating patient to stop smoking
  Statins prescribed
  Rate of catheter related UTI
  Rate of aspiration pneumonia
  Hospital length of stay
  Discharge destination
  The time frame for this project is 5 years. All elements of acute stroke care will be collected during the hospital stay.

SECONDARY OUTCOMES:
To assess the rate of antiplatelet agent used for stroke prevention. | 5 years
  This would include the rate of patients being prescribed dual antiplatelet therapy, and the duration/compliance of taking antiplatelet medicine.
To assess the rate of using anticoagulant medication for stroke prevention in patients with atrial fibrillation. | 5 years
  To assess the rate of bridging therapy used during hospitalization. Bridging therapy is to give intravenous or subcutaneous anticoagulation while waiting for warfarin to be therapeutic. In addition, the rate of prescribing new oral anticoagulants for stroke prevention in atrial fibrillation will be assessed,

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Dong, M.D., Ph.D, Principal Investigator — Shanghai Stroke Service System
Locations (11):
- China (11):
  - Zhongshan Hospital affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Huashan Hospital，Fudan University, Shanghai, Shanghai Municipality
  - Shuguang Hospital affiliated to Shanghai Traditional Chinese Medicine University, Shanghai, Shanghai Municipality
  - The Shanghai Tenth People's Hospital, Tongji University, Shanghai, Shanghai Municipality
  - Dongfang Hospital affiliated to Shanghai University of TCM, Shanghai, Shanghai Municipality
  - Renji hospital，Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Changhai Hospital, Shanghai, Shanghai Municipality
  - Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality
  - Shanghai Jiao Tong University School of Medicine Ruijin Hospital, Shanghai, Shanghai Municipality
  - Shanghai Ninth People's Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - The Sixth People's Hospital affiliated to Shanghai Jiaotong University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Yes
The data is planning to make individual participant data available, especially to anticipating collaborator.

REFERENCES:
- [Derived] Xu J, Xie Y, Fang K, Wang X, Chen S, Liu X, Zhao Y, Guan Y, Cai D, Li G, Liu J, Liu J, Zhuang J, Xian Y, Shen H, Li H, Wang DZ, Campbell BC, Parsons MW, Dong Y, Dong Q. Effect of the Shanghai Stroke Service System (4S) on the quality of stroke care and outcomes: A prospective quality improvement project. Int J Stroke. 2023 Jun;18(5):599-606. doi: 10.1177/17474930221125993. Epub 2022 Oct 15. PMID 36082948
- [Derived] Dong Y, Han Y, Shen H, Wang Y, Ma F, Li H, Wang Y, Dong Q. Who may benefit from lower dosages of intravenous tissue plasminogen activator? Results from a cluster data analysis. Stroke Vasc Neurol. 2020 Dec;5(4):348-352. doi: 10.1136/svn-2020-000388. Epub 2020 Jul 1. PMID 32611728
- [Derived] Dong Y, Fang K, Wang X, Chen S, Liu X, Zhao Y, Guan Y, Cai D, Li G, Liu J, Liu J, Zhuang J, Wang P, Chen X, Shen H, Wang DZ, Xian Y, Feng W, Campbell BC, Parsons M, Dong Q. The network of Shanghai Stroke Service System (4S): A public health-care web-based database using automatic extraction of electronic medical records. Int J Stroke. 2018 Jul;13(5):539-544. doi: 10.1177/1747493018765492. Epub 2018 Mar 21. PMID 29561219